CLINICAL TRIAL: NCT02905318
Title: A Phase II Study of Palbociclib, A CDK4/6 Inhibitor, in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Palbociclib in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I223
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbociclib (Experimental): 125mg orally days 1-21 every 28 day cycle
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — 125 mg orally on days 1-21 each 28 day cycle

SUMMARY:
The purpose of this study is to find out what effects a new drug, palbociclib, has on prostate cancer and will look at the side effects of treatment with palbociclib. The researchers doing this study are also interested in looking for markers that may help predict which patients are most likely to be helped by palbociclib and to see how the cancer cells respond to palbociclib.

DETAILED DESCRIPTION:
The standard or usual treatment for this disease may be chemotherapy or other types of treatment to slow the spread of the disease and relieve some symptoms of cancer.

Palbociclib is a new type of drug for prostate cancer. Laboratory tests show that it may help slow the growth of prostate cancer. Palbociclib has been shown to help patients with breast cancer but it is not known if the drug is useful for treating prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed adenocarcinoma of the prostate without evidence of small cell/neuroendocrine differentiation.
* Patients must consent to blood collection for testing prior to enrollment by a central reference laboratory. Screening will be done through the CRPC Master Screening Protocol (IND234)
* Patients must have clinically and/or radiologically documented disease. Patients with elevated PSA only are not eligible. All radiology studies must be performed within 28 days prior to enrollment (within 35 days if negative).
* All patients must have consented to the release of a tumour block from their primary or metastatic tumour. The centre/pathologist must have agreed to the submission of the specimen.
* Patients must have evidence of either biochemical or radiological disease progression in the setting of surgical or medical castration:

  * PSA progression:

    * Minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement
    * PSA must be ≥2.0 ug/L
  * Objective progression:

    * RECIST 1.1 or
    * Soft tissue or visceral disease progression or
    * PCWG3 for bone progression (>2 new lesions on bone scan or CT)
  * Surgical/medical castration:

    * Prior orchiectomy or
    * LHRH agonist/antagonist and testosterone < 50 ng/dL or < 1.7 nmol/L. LHRH agonist/antagonist therapy must be maintained for the duration of study therapy and if previously discontinued, must be restarted and castrate level of testosterone present.
* Patients must be ≥18 years of age.
* ECOG performance status 0 or 1 (Appendix I) and have a life expectancy of ≥ 6 months.
* Previous Therapy:

Patients must have recovered from any treatment-related toxicities prior to registration (unless ≤ grade 1, irreversible, or considered by investigator as not clinically significant).

Surgery:

Prior major surgery is permitted provided that a minimum of 14 days have elapsed between any major surgery and enrollment (7 days for minor surgery e.g. port insertion), and that wound healing has occurred.

Radiation:

Prior external beam radiation or radium-223 is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose and enrollment. Limited field radiation (for example less than 25% of marrow bearing bones) for palliation of bone pain is permitted < 2 weeks prior to starting study drug. Concurrent radiation is not permitted. Prior strontium-89 at any time is not permitted.

Systemic Therapy:

Prior systemic therapy is permitted as outlined below. Patients must have recovered from all reversible toxicity related to prior systemic therapy and have adequate washout prior to enrollmentas follows and as specified in the Sections below:

Longest of one of the following:

* Two weeks;
* The longer of 30 days or 5 half-lives for investigational agents;
* Standard cycle length of standard therapies.

Hormonal Therapy: Patients must have received prior hormonal treatment with at least one of abiraterone acetate, enzalutamide, ARN-509 TAK-700 and TOK-001. Prior anti-androgen therapy must have been discontinued at least 28 days (or 42 days for bicalutamide) prior to enrollment.

Cytotoxic Therapy: Patients may have received docetaxel therapy in the castrate sensitive setting as well as up to 1 regimen of any cytotoxic therapy in the CRPC setting. Prior treatment with docetaxel, cabazitaxel and mitoxantrone is permitted.

Immunotherapy: Patients may have received prior immune checkpoint inhibitors (anti PDL1 and anti CTL-4); vaccines and treatment with oncolytic viruses is permissible.

Other therapy:

* Previous therapy with CDK or mTOR inhibitors is not allowed.
* Prior treatment with other agents, such as tyrosine kinase or other targeted agents is permissible.
* Systemic corticosteroids are permitted at a dose equivalent to <10 mg prednisone daily; topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are permitted.
* Bisphosphonates / denosumab are permitted for treatment of hypercalcemia, osteoporosis and skeletal-related events.

  * Laboratory Requirements (within 7 days of enrollment):

Neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Hemoglobin ≥ 100 g/L Bilirubin ≤ 1.5 x ULN; if confirmed Gilbert's then bilirubin ≤ 3.0 x ULN AST and ALT ≤ 1.5 x ULN; if patient has liver metastases ≤ 5.0 x ULN Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥ 50 mL/min;

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient enrollment.
* Men of childbearing potential must have agreed to use a highly effective contraceptive method during treatment and for 90 days after stopping treatment and should not father a child or donate sperm during this period.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Patients with central nervous system (CNS) involvement unless at least 4 weeks from prior therapy completion (including radiation and/or surgery) AND clinically stable and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
* Patients with serious illnesses or medical conditions which could cause unacceptable safety risks or would not permit the patient to be managed according to the protocol. This includes but is not limited to:

  * active infection requiring systemic therapy;
  * uncontrolled/severe cardiovascular disease
  * active or known human immunodeficiency virus (HIV);
* Patients who are unable to swallow oral medication and/or have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients with history of hypersensitivity to palbociclib or any of its excipients.
* Patients who have been treated with prior CDK4/6 inhibitors, mTOR inhibitors or strontium-89 at any time or require continued or concurrent treatment with:

  * Systemic corticosteroids at a dose equivalent to prednisone > 10 mg daily. Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed.
  * Any medications or substances that are potent/strong inhibitors or inducers of CYP3A isoenzymes. All patients must have discontinued these medications at least 7 days prior to the first dose of protocol treatment (at least 14 days for herbal/dietary supplements and traditional Chinese medicines).
  * Bisphosphonates / denosumab for reasons other than hypercalcemia, osteoporosis or skeletal-related events.
  * Warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), factor X inhibitors or fondaparinux is allowed.
  * Other anti-cancer or investigational agents (except LHRH)
* Patients with a history of non-compliance to medical regimens.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate estimated by proportion of evaluable patients who had CR, PR or SD as their best response to treatment | 36 months
  Clinical benefit is defined as one of the following:
  * PSA decline ≥ 50%
  * CR or PR (objective)
  * SD for ≥12 weeks (objective, without PSA progression)

SECONDARY OUTCOMES:
Effect of Palbociclib on PSA decline based on decrease in PSA test values from the baseline value | 36 months
Objective response determined by RECIST 1.1 | 36 months
Progression-free survival | 36 months
Overall survival | 36 months
Number and severity of adverse events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim Chi, Study Chair — BCCA - Vancouver Cancer Centre, BC Canada
Locations (7):
- Canada (7):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No